CLINICAL TRIAL: NCT02153931
Title: Effects of an Internet Support Group for Parents of a Child With Neurofibromatosis Type 1
Brief Title: Internet Support Group for Parents of a Child With Neurofibromatosis Type 1
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140113; 14-C-0113
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01-29

CONDITIONS: Neurofibromatosis 1
Keywords: Children's Tumor Foundation; Social Support; Online; Anxiety; Depression
MeSH Terms: conditions — Neurofibromatosis 1; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Volunteers: Parents of children with NF1

SUMMARY:
Background:

- Studies show that Internet Support Groups (ISGs) can help parents of children with chronic conditions. Researchers want to find out if ISGs can help parents of a child with the genetic disorder Neurofibromatosis Type 1 (NF1).

Objective:

- To see if an ISG for parents with a child with NF1 can give the parents more social support and less anxiety.

Eligibility:

- Adults age 18 and older with a child (age 0 25 years) with NF1.

Design:

* Participants will register for the study on a website hosted by the Children s Tumor Foundation.
* Participants will complete 5 questionnaires. These will be about their emotional well-being, their child s health status, and their contact information.
* The ISG will include a Discussion Forum that participants can enter 24 hours a day, 7 days a week. A professional moderator will post questions and discussion topics. The moderator can also respond to questions. They will be a psychologist, a psychology associate, or a nurse-practitioner. Each one will be highly experienced at working with young people with NF1 and their families.
* The ISG also will contain a chat room. Here participants can chat with other users in real time. The chat room will be open for one 90-minute session per week.
* The ISG will remain open for 8 weeks. Then participants will retake 4 of the questionnaires from the beginning of the study. They will also complete 1 other questionnaire about their experiences with the ISG. Information from any messages participants post on the ISG website will be collected.
* Three months after the ISG closes, participants will complete the questionnaires one final time.

DETAILED DESCRIPTION:
BACKGROUND:

* The complex symptom profile in NF1 puts children and adolescents with this condition at risk for a variety of physical, cognitive, and social-emotional difficulties. Thus, caring for a child with a chronic medical condition such as NF1 can be challenging.
* Over the last two decades, researchers have been examining the use of internet support groups (ISGs) as a means of connecting individuals with similar conditions, diagnoses, or challenges to provide emotional and informational support.
* While the benefits of ISGs have been well documented in many studies of medical patients, very few have examined the use of ISGs in parents of children with chronic medical conditions. Further, no studies have been conducted on an ISG in parents of a child with NF1.

OBJECTIVES:

* The primary objective of this pilot study is to assess the effectiveness of an ISG designed for parents of children with NF1 on a measure of perceived social support.
* Secondary objectives are to assess effects of the ISG on self-efficacy, depression, and anxiety, and to explore themes and topics discussed in the ISG.

ELIGIBILITY:

Eligible participants must self-report:

* Being greater than or equal to 18 years of age
* Having a child with a diagnosis of NF1 between 0 and 25 years of age
* Living in the same home as the child with NF1

  * Having regular access to a computer with internet capability

DESIGN:

* Parents of children with NF1 will be recruited through Dr. Widemann s NF1 patient database and through the Children s Tumor Foundation s (CTF) NF registry.
* Eligible participants will be emailed a link to access the study website through the CTF website. Due to the nature of the study, consent will be obtained online.
* After consenting, participants will be administered (electronically) baseline measures of perceived social support, self-efficacy, depression, and anxiety. After 8 weeks, participants will complete the measures again via the same website, as well as a post-study questionnaire assessing their experiences with participation. Measures will be repeated at 3-months post-intervention.
* Content analyses will be performed to identify themes and needs of the participants

ELIGIBILITY:
* ELIGIBILITY CRITERIA

INCLUSION CRITERIA FOR PARENT PARTICPANT:

Participants must self-report being the primary caregiver of one or more children ages 0 to 25 with a confirmed diagnosis of NF1.

Participants must report being at least 18 years of age.

Participants must report living in the same home as the child(ren) with NF1 a majority of the time.

Participants must report having regular access to a computer and internet connection.

Participants will indicate they do not have any plans to start any other internet support group for parents of children with NF during the study time period.

Participants must have the ability to read and communicate in the English language.

Participants must have the ability to understand and the willingness to provide an online informed consent document.

EXCLUSION CRITERIA FOR PARENT PARTICIPANT:

Although individuals will be allowed to participate if they currently are part of another internet forum for NF, they will be excluded if they report they plan to start a new internet support group during the study period.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-05-31; Primary Completion 2015-04-06 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
ISG effects on perceived support | 3 months
  To determine the effects of an ISG on perceived social support among parents of a child with NF1 from baseline to 8 weeks and frombaseline to 3 months postintervention.

SECONDARY OUTCOMES:
ISG effects on depression and anxiety | 3 months
  To determine the effects of an ISG on perceived social support among parents of a child with NF1 from baseline to 8 weeks and frombaseline to 3 months post-intervention.
Identify themes and needs of chat room support | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Staci M Peron, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States